CLINICAL TRIAL: NCT06146543
Title: Stress Ball During Lumbar Puncture in Neurological Patients the Effect of the Application on Anxiety Level
Brief Title: Stress Ball During Lumbar Puncture the Effect of the Application on Anxiety Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Dilek Baykal, Assistant Professor, Atlas University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2135111
Record Dates: First submitted 2023-11-11; First posted 2023-11-24 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neurology patients (Experimental): Patients coming to the neurology clinic for lumbar puncture.
  Interventions: Other: Stress ball
- Control (No Intervention): The scale will be applied to the same patient group before and after lumbar puncture without intervention.

INTERVENTIONS:
Other: Stress ball — Before the procedure begins, the patient's free hand will be given an elastic ball that is large enough to hold in the palm of the hand and squeeze easily. He/she will be asked to squeeze this ball slowly throughout the process. At the end of the procedure, the ball will be removed from his hand and the patient will be relieved.
  Arms: neurology patients

SUMMARY:
Individuals who come to the neurology clinic to undergo lumbar puncture, and meet the inclusion criteria, and agree to participate in the study will be given a stress ball during the procedure and will be asked to squeeze this ball.

DETAILED DESCRIPTION:
Before starting the research, the purpose of the research will be explained to patients who meet the inclusion and exclusion criteria, and their verbal and written consent will be obtained. The Declaration of Helsinki will be adhered to throughout the research. Data will be obtained by administering face-to-face surveys. The population of the study will be individuals who meet the inclusion criteria at the neurology clinic of Istanbul University - Istanbul Faculty of Medicine, and the individuals who agree to participate in the study will constitute the sample. To determine the number of samples, a comparison of two groups was made using the "G-Power 3.1.7" program. The minimum sample size that would provide Type I margin of error (α): 0.05 and power of the test (1-β): 0.80 was determined as 47 people in total. Taking into account sample loss, it was aimed to reach a total of 50 people.

Then, the form questioning socio-demographic information and the STAI XT State-Trait Anxiety Scale will be applied. Before the LP begins, the patient's free hand will be given an elastic ball that is large enough to hold in the palm of the hand and squeeze easily. He/she will be asked to squeeze this ball slowly throughout the process. At the end of the procedure, the ball will be removed from his hand and the patient will be relieved. After the patient is relaxed, the STAI XT State-Trait Anxiety Scale will be administered again.

The state anxiety scale is a sensitive scale for evaluating sudden changes in emotional reactions. The trait anxiety scale aims to measure the continuity of anxiety that a person generally tends to experience. Since this study aims to evaluate the anxiety levels of patients regarding their current situations, the state anxiety scale will be used.

ELIGIBILITY:
Inclusion Criteria:

* -Being over 18 years old
* Volunteering to participate in the study
* Being able to read and write
* No problems in verbal communication
* Lumbar puncture procedure will be performed

Exclusion Criteria:

* - Do not come to the neurology clinic for any procedure other than lumbar puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
STAI XT-1 State-Trait Anxiety Scale | up to 6 months
  It will be used to evaluate the current state of anxiety. The scale has a total of 40 items, 20 of which measure state anxiety and 20 measure trait anxiety. In order to determine the behaviors and emotions of the individuals to whom the scale is applied, each item is evaluated with the options of 'not at all', 'somewhat', 'a lot', and 'completely'. An increase in the total score obtained from the scale indicates that the person's anxiety level is increasing.
  When the patient comes to the clinic, he/she will be informed about the study his/her consent will be obtained, and then the scale will be filled out.

SECONDARY OUTCOMES:
STAI XT-1 State-Trait Anxiety Scale | up to 6 months
  It will be used to evaluate the immediate anxiety state after the intervention. The scale has a total of 40 items, 20 of which measure state anxiety and 20 measure trait anxiety. In order to determine the behaviors and emotions of the individuals to whom the scale is applied, each item is evaluated with the options of 'not at all', 'somewhat', 'a lot', and 'completely'. An increase in the total score obtained from the scale indicates that the person's anxiety level is increasing.
  After the lumbar puncture procedure is completed, the patient will be relieved by taking the ball from her hand and the scale will be filled.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No